CLINICAL TRIAL: NCT01333449
Title: Prospective Phase II Study of Decitabine Induction Therapy to Reduce Pre-transplant Disease Burden Prior to Allogeneic Hematopoietic Cell Transplant in Patients With Newly Diagnosed Myelodysplastic Syndromes.
Brief Title: Study of Decitabine Induction Prior to Allogeneic Hematopoietic Cell Transplant in Newly Diagnosed MDS Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor subject accrual
Sponsor: Singapore General Hospital (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Decitabine01
Record Dates: First submitted 2010-11-30; First posted 2011-04-12 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Myelodysplastic Syndrome
Keywords: Decitabine; MDS, myelodysplastic syndrome; prospective open label, phaseII; Allogeneic Hematopoietic cell transplant
MeSH Terms: conditions — Myelodysplastic Syndromes; Anemia, Refractory, with Excess of Blasts | interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental): Decitabine 20mg/m^2 infusion one hour per day, for 5days,every 28days,total 2-6cycles.
  Interventions: Drug: Decitabine

INTERVENTIONS:
Drug: Decitabine — 20mg/m^2 infusion one hour per day, for 5days,every 28days,total 2-6cycles.
  Other Names: Dacogen

SUMMARY:
Allogeneic blood stem cell transplant remains the only potential curative treatment for myelodysplastic syndromes (MDS) to date. Pre-transplant induction chemotherapy with leukemia-type regimens is associated with significant toxicity and even death. The hypomethylating agents decitabine and 5-azacytidine have been shown in studies to cause improved hematologic parameters and partial or complete responses in patients with high risk MDS compared to standard therapy. In contrast to leukemia-type chemotherapy, decitabine is associated with a relatively low risk of toxicity. We therefore propose to treat transplant-eligible MDS patients with Decitabine as induction therapy and a bridge to transplant.

Hypothesis:

1. Decitabine is able to reduce disease burden as measured by blood and marrow blast counts prior to allogeneic hematopoietic stem cell transplant to below 5%.
2. Decitabine is well-tolerated by patients with high-risk MDS and will be a safe induction agent and bridge prior to allogeneic transplant in transplant-eligible patients.

DETAILED DESCRIPTION:
Primary endpoint:

1. safety and tolerability of Decitabine prior to transplant (assessed by occurence of non-hematologic toxicities of grade 3 or more as defined by CTC grading)
2. reduction in pre-transplant disease burden ability to achieve blast <5% in the bone marrow and peripheral blood

Secondary endpoints:

1. Proportion of patients with suitable donor able to proceed to an allogeneic hematopoietic cell transplant.
2. Non-relapse mortality
3. time to neutrophil engraftment
4. Overall survival and disease-free survival.

Patients will receive Decitabine until blast <5% is achieved, suitable HLA-matched donor or umbilical cord blood is available up to a maximum of 6 cycles. Patient who progress on therapy or are unable to find a donor by 6 cycles will be removed from protocol. The method, conditioning regimen and choice of donor will be determined based on patient's age and functional status, and transplant physician's discretion. The available regimens are standardized within the center

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed MDS patients aged 21 to 65 years belonging to any of the following categories: refractory cytopenia with multilineage dysplasia (RCMD) with or without ringed sideroblasts (i.e. RCMD and RCMD-RS), refractory anemia with excess blasts-1 (RAEB-1) or RAEB-2 if the prognostic scores are IPSS (international prognostic scoring system) Int-2 or IPSS-high or with WPSS (WHO prognostic scoring system) 3 and above
2. Therapy-related MDS with IPSS Int-2 and above or WPSS 3
3. Acceptable cardiac function MUGA or Echocardiography left ventricular ejection fraction of 40% and above
4. Acceptable lung function: FEV1>70% predicted, DLCO>60% predicted
5. Acceptable renal function: CCT > 50ml/min
6. Acceptable liver function: abnormalities in bilirubin or transaminases not > 2times upper limit of normal
7. Performance status of ECOG 2 or HCT-specific Comorbidity Index < 3

Exclusion Criteria:

1. Any co-morbidity other than MDS which limits life-expectancy to <3mth
2. Diagnosis of other active cancer other than squamous cell carcinoma, basal cell carcinoma or carcinoma-in-situ 1 or 2 of the cervix
3. Presence of active infections not under control
4. Receipt of 5-azacytidine or other induction chemotherapy for MDS/AML
5. Patients not keen to explore allogeneic HCT as part of curative treatment plan
6. Pregnancy

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-07; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Reduction in pre-transplant disease burden | 2 years

SECONDARY OUTCOMES:
Proportion of patients with suitable donor able to proceed to an allogeneic HCT | 2 years
Non-relapse mortality | 3 years
Time to neutrophil engraftment | 2 years
Overall survival survival | 3 years
Disease free survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Aloysius Ho, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore, Singapore